CLINICAL TRIAL: NCT05942729
Title: Etiological DiagnOsis of caRdiac Diseases Based on echoCardiograpHIc Images and Clinical Data.
Acronym: ORCHID
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0819
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hypertension Arterial; Hypokinetic; Cardiomyopathies; Left Ventricular Hypertrophy
Keywords: Hypertension; HTN; Arterial Hypertension; Artificial Intelligence; AI; Cardiac remodelling; Left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Sedentary Behavior; Cardiomyopathies; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hypokinetic cardiomyopathy.: The first arm includes patients with hypokinetic cardiomyopathy for whom echocardiographic data do not readily distinguish between a cause related to coronary artery disease or related to primary myocardial dysfunction, requiring invasive intervention, i.e., coronary angiography.
  Interventions: Other: Determine the etiology of hypokinetic and hypertrophic heart disease on transthoracic echocardiography data alone
- Patients with left ventricular hypertrophy related to hypertension/infiltrative myocardial disease: The second arm includes patients with left ventricular hypertrophy, whose aetiology may be various and whose workup is particularly extensive and expensive.
  Interventions: Other: Determine the etiology of hypokinetic and hypertrophic heart disease on transthoracic echocardiography data alone

INTERVENTIONS:
Other: Determine the etiology of hypokinetic and hypertrophic heart disease on transthoracic echocardiography data alone — The origin of the pathology will have been previously diagnosed for each patient thanks to complementary examinations performed as part of routine care (e.g. cardiac CT, cardiac MRI, coronary angiography, thorough biology, nuclear medicine). This information will be used (i) to guide the learning of the AI method developed during the project from a sub-population (80% of the collected database will be used to train the algorithms); (ii) to serve as an evaluation criterion from a test sub-population (remaining 20% of the collected database)

SUMMARY:
Research hypothesis - Recent studies have shown that high-dimensional descriptors of the cardiac function can be efficiently exploited to characterize targeted pathologies. In this project, the investigators hypothesize that echocardiograms possess a wealth of information that is currently under-exploited and that, combined with relevant patient data, will allow the development of robust and accurate digital tools for etiological diagnosis.

Objectives - Based on key advances recently obtained in image analysis, notably by members of the consortium, the objective of this project is to develop rigorous and explainable cardiac disease prediction models from echocardiography based on the transformer paradigm (AI). The strength of this study lies in the development of a strong AI framework to model the complex interactions between high-quality image-based measurements extracted from echocardiograms and relevant patient data to automatically predict etiological diagnosis of cardiac diseases

ELIGIBILITY:
Inclusion Criteria:

* Patients with transthoracic echocardiography with satisfactory image quality (sufficient echogenicity)

Exclusion Criteria:

* Minor patients
* Patients under curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two distinct populations are targeted in this project. The first concerns patients with hypokinetic cardiomyopathy for whom echocardiographic data do not easily distinguish between a cause related to coronary artery disease or related to primary myocardial dysfunction, imposing the performance of an invasive intervention, i.e., a coronary angiography. The second concerns patients with left ventricular hypertrophy, whose etiology can be diverse and whose assessment is particularly exhaustive and costly. In this project, we will study the two most frequent causes: arterial hypertension and infiltrative myocardial disease. The cohort will be composed in a balanced way with respect to the four pathologies mentioned above as well as through data from patients without significant heart disease. This database will be constructed from patients who have been hospitalized at the Cardiology Department during the period January 2018 to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
the comparison of the performance of the etiological diagnosis obtained by the artificial intelligence with the etiological diagnosis already established and validated by a physician from the complementary examinations performed on the targeted patients. | Baseline
  The origin of the pathology being previously diagnosed for each patient thanks to complementary examinations carried out in routine (e.g.: cardiac scanner, cardiac MRI, coronary angiography, thorough biology, nuclear medicine). This information will be used (i) to guide the learning of the AI method developed during the project from a sub-population (80% of the collected database will be used to train the algorithms); (ii) to serve as an evaluation criterion from a test sub-population (remaining 20% of the collected database). In addition, visualization tools will be developed to allow clinicians to analyze and interpret the results, particularly with respect to the decision mechanism performed by the algorithm to predict the origin of the pathology. In particular, attention maps will be displayed that will simply allow clinicians to see which data or part of the data was assembled in order to make the decision.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lyon Sud, Pierre-Bénite, France